CLINICAL TRIAL: NCT00000114
Title: Randomized Trial of Vitamin A and Vitamin E Supplementation for Retinitis Pigmentosa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: NEI-10
Record Dates: First submitted 1999-09-23; First posted 1999-09-24 (Estimated); Last update posted 2009-09-17 (Estimated); Status verified 2009-09

CONDITIONS: Retinitis Pigmentosa
Keywords: retinitis pigmentosa; vitamin supplements
MeSH Terms: conditions — Retinitis Pigmentosa | interventions — Vitamin E; Vitamin A

INTERVENTIONS:
Drug: Vitamin E
Drug: Vitamin A

SUMMARY:
To determine whether supplements of vitamin A or vitamin E alone or in combination affect the course of retinitis pigmentosa.

DETAILED DESCRIPTION:
Retinitis pigmentosa (RP) is a group of inherited retinal degenerations with a worldwide prevalence of about 1 in 4,000. Patients typically report night blindness in adolescence and lose vision in the midperipheral followed by far-peripheral visual field in adulthood due to progressive loss of both rod and cone function. Most patients have reductions in central vision by age 50 to 80 years. Modern-day electroretinograms (ERGs) make it possible to record retinal responses from most patients with remaining vision and thereby monitor objectively the course of their disease.

While the natural course of retinal degeneration in the common forms of RP was being studied, it was noted that a subgroup of patients aged 18 through 49 who were treating themselves with both vitamin A and vitamin E and other nutritional supplements exhibited less decline in ERG amplitude over a 2-year period. These preliminary findings, as well as the known roles of vitamins A and E in maintaining normal photoreceptor function and structure, prompted this randomized, controlled trial to determine whether these vitamins alone or in combination would halt or slow the progression of the common forms of RP.

This study was a randomized, controlled double-masked trial with 2 x 2 factorial design and duration of 4 to 6 years. Patients were assigned to one of four treatment groups:

15,000 IU/day vitamin A

15,000 IU/day vitamin A + 400 IU/day vitamin E

trace amounts of both vitamins A and E

400 IU/day of vitamin E

The main outcome measure was the 30-Hz cone ERG amplitude. In addition, visual field and visual acuity were measured annually.

ELIGIBILITY:
Men and nonpregnant women between ages 18 and 49 years with common forms of RP were included. All eligible patients had retinal arteriolar attenuation, elevated dark adaptation thresholds, and reduced ERGs. Patients had best corrected Snellen visual acuity of 20/100 or better, central visual field diameter on the Goldman perimeter with V4 e white test light of 8 degrees or greater, and ERG amplitude of 2.5 or greater in response to 0.5-Hz white light or of 0.12 ultraviolet light or greater in response to 30-Hz white flickering light in at least one eye. In addition, patients had normal fasting serum retinol and serum liver function profile and weight above the lower fifth percentile for age, sex, and height. All patients had a total estimated pre-trial intake of vitamins A and E from diet plus pills not greater than 11,500 IU/day and 40 IU/day, respectively.

Ages: 18 Years to 49 Years | Sex: All
Age Groups: Adult
Dates: Start 1984-05; Study Completion 1987-06 (Actual)

REFERENCES:
- [Background] Berson EL, Rosner B, Sandberg MA, Hayes KC, Nicholson BW, Weigel-DiFranco C, Willett W. A randomized trial of vitamin A and vitamin E supplementation for retinitis pigmentosa. Arch Ophthalmol. 1993 Jun;111(6):761-72. doi: 10.1001/archopht.1993.01090060049022. PMID 8512476
- [Background] Sandberg MA, Weigel-DiFranco C, Rosner B, Berson EL. The relationship between visual field size and electroretinogram amplitude in retinitis pigmentosa. Invest Ophthalmol Vis Sci. 1996 Jul;37(8):1693-8. PMID 8675413
- [Derived] Comander J, Weigel DiFranco C, Sanderson K, Place E, Maher M, Zampaglione E, Zhao Y, Huckfeldt RM, Bujakowska KM, Pierce E. Natural history of retinitis pigmentosa based on genotype, vitamin A/E supplementation, and an electroretinogram biomarker. JCI Insight. 2023 Aug 8;8(15):e167546. doi: 10.1172/jci.insight.167546. PMID 37261916